CLINICAL TRIAL: NCT07272512
Title: Prospective Multicenter Real-world Study of Surufatinib in Patients With Advanced Neuroendocrine Neoplasms
Acronym: ZSPAC-17
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-NEN116
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Neoplasms
Keywords: surufatinib; advanced neuroendocrine tumors; advanced neuroendocrine neoplasms
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — surufatinib

STUDY DESIGN:
Intervention Model Description: Prospective multicenter phase 4, single-group assignment, open-label study of surufatinib in patients with advanced neuroendocrine neoplasms
Masking Description: This is an open-label study; no masking is implemented for any study personnel or participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib Treatment (Experimental): Adult patients with histologically or cytologically confirmed advanced neuroendocrine neoplasms (NENs) will receive oral surufatinib according to routine clinical practice and protocol guidance. Surufatinib will be administered either as monotherapy (300 mg once daily in continuous 4-week cycles) or as part of combination therapy (250 mg once daily) at the discretion of the treating physician. Treatment will continue until radiologic or clinical disease progression, unacceptable toxicity, withdrawal of consent, death, or end of study, whichever occurs first. Concomitant anticancer therapies, dose modifications, and interruptions are permitted and will be managed in accordance with the protocol and local standard of care.
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib (Sulanda, HMPL-012) is an oral small-molecule tyrosine kinase inhibitor that selectively targets VEGFR1-3, FGFR1 and CSF1R, exerting both anti-angiogenic and immune-modulating effects. In this study, surufatinib will be administered as film-coated tablets once daily: 300 mg QD for monotherapy or 250 mg QD when used in combination regimens, according to protocol guidance and the treating physician's judgment. Treatment is given in continuous 4-week cycles and continued until disease progression, unacceptable toxicity, withdrawal of consent, death, or end of study. Dose interruptions and reductions are allowed and will be managed following the protocol and the approved prescribing information.

SUMMARY:
This is a prospective, multicenter, phase 4, single-arm study designed to evaluate the effectiveness and safety of surufatinib in adult patients with advanced neuroendocrine neoplasms (NENs) treated in routine clinical practice. Approximately 350 patients with histologically or cytologically confirmed advanced NENs and at least one measurable lesion (RECIST 1.1) will receive oral surufatinib, either as monotherapy (300 mg once daily in 4-week cycles) or in combination regimens (250 mg once daily), according to the treating physician's judgment and protocol guidance.

Participants will be followed with regular imaging, laboratory tests, cardiac assessments, and patient-reported outcome questionnaires to monitor tumor response, side effects, quality of life, and treatment adherence. The primary outcomes include progression-free survival, objective response rate, disease control rate, and overall survival; safety will be assessed by the type, frequency, and severity of adverse events. The findings are expected to inform standardized, evidence-based use of surufatinib and help optimize individualized treatment strategies for patients with advanced NENs in the real-world setting.

DETAILED DESCRIPTION:
This is a prospective, multicenter, phase 4, single-arm, open-label study designed to systematically characterize the real-world use of surufatinib in adult patients with advanced neuroendocrine neoplasms (NENs). Surufatinib is an oral small-molecule tyrosine kinase inhibitor with dual antitumor activity through anti-angiogenic and immune-modulating mechanisms, and has shown clinically meaningful efficacy in phase 3 trials in both pancreatic and extra-pancreatic NETs. However, evidence is still limited regarding its effectiveness, safety profile, patterns of use (monotherapy versus combination regimens, line of therapy, cross-line use), and impact on quality of life in routine clinical practice in China.

Approximately 350 patients with histologically or cytologically confirmed advanced NENs and at least one measurable lesion (RECIST 1.1) will be enrolled from multiple centers. According to the treating physician's judgment and protocol guidance, patients will receive oral surufatinib either as monotherapy (300 mg once daily in 4-week cycles) or in combination regimens (250 mg once daily), and treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, death, or end of study. Tumor assessments, laboratory tests, cardiac monitoring, and patient-reported outcome questionnaires (including generic and NET-specific quality-of-life scales and a medication-adherence scale) will be performed at regular intervals during follow-up. The study will estimate progression-free survival, objective response rate, disease control rate, and overall survival, describe the incidence and severity of treatment-emergent adverse events, and explore how baseline clinicopathological features and treatment patterns are associated with outcomes, with the aim of developing evidence-based, standardized, and individualized clinical pathways for the real-world use of surufatinib in advanced NENs.

ELIGIBILITY:
Inclusion Criteria:

* Adequately understand the study and voluntarily sign the Informed Consent Form.
* Have a confirmed histological or cytological diagnosis of neuroendocrine neoplasm.
* Have measurable disease based on RECIST 1.1.
* Have adequate organ and bone marrow function.
* Life expectancy > 12 weeks.
* Women of childbearing age must be willing to use adequate contraceptives during the study period of drug treatment.

Exclusion Criteria:

* Other malignant tumors diagnosed within 5 years (excluding effectively treated basal cell carcinoma, cutaneous squamous cell carcinoma, or completely resected in situ cervical/breast cancer).
* Concurrent use of other investigational drugs or approved/investigational anti-tumor therapies.
* Contraindications to surufatinib: active bleeding, ulcers, intestinal perforation/obstruction, uncontrolled hypertension, grade III-IV cardiac insufficiency, <30 days post-major surgery, or severe hepatic/renal impairment.
* Pregnant (positive pre-treatment pregnancy test) or lactating females.
* Massive pleural effusion/ascites requiring drainage.
* Other diseases/abnormalities (metabolic, physical, or laboratory) deemed by the investigator to preclude study drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-11-29 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 12 months
  From the date of enrollment to the date of the first onset of disease progression or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate (DCR) | up to 12 months
  CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Overall survival (OS) | up to 36 months
  From the date of enrollment to the date of the first onset of death from any cause

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital shanghai jiao tong university school of medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No